CLINICAL TRIAL: NCT07156097
Title: Comparative Effects of a Boron-Enriched Diet and a Mediterranean-Style Diet on Gut Microbiota, Appetite-Regulating Hormones, and Cardiometabolic Parameters in Obese Adults: A Controlled Intervention Study
Brief Title: Effects of Boron and Mediterranean Diets on Gut Microbiota and Metabolic Health
Acronym: BOR-SAFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Feray ÇAĞIRAN YILMAZ, Associate Professor, Dicle University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/01-19
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Dietary Intervention; Gut Microbiota; Cardiometabolic Risk Factors; Appetite-Regulating Hormones
Keywords: Boron-enriched diet; Mediterranean diet; gut microbiota; obesity; cardiometabolic health; Appetite hormones
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups: a boron-rich diet group or a Mediterranean-style diet group. Each intervention was applied for 4 weeks, and outcomes related to obesity, microbiota, cardiometabolic risk markers, and appetite-regulating hormones were assessed
Masking Description: No masking was applied. Both participants and investigators were aware of the dietary intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boron-rich Diet (Experimental): Participants followed a 4-week dietary intervention emphasizing boron-rich foods (e.g., legumes, nuts, dried fruits). The aim was to assess effects on obesity, microbiota composition, appetite hormones, and cardiometabolic risk markers.
  Interventions: Other: Boron-rich Diet
- Mediterranean-style Diet (SAFF) (Active Comparator): Participants followed a 4-week Mediterranean-style dietary pattern (SAFF), characterized by high intake of vegetables, fruits, whole grains, olive oil, and lean protein sources. This arm served as a comparator for the boron-rich diet.
  Interventions: Other: Mediterranean-style Diet (SAFF)

INTERVENTIONS:
Other: Mediterranean-style Diet (SAFF) — Participants followed a 4-week Mediterranean-style dietary pattern (SAFF), characterized by high intake of vegetables, fruits, whole grains, olive oil, and lean protein sources. This arm served as a comparator for the boron-rich diet.
  Arms: Mediterranean-style Diet (SAFF)
Other: Boron-rich Diet — Participants assigned to this arm will follow a boron-rich dietary pattern for 4 weeks. The diet includes foods naturally high in boron (e.g., dried fruits, nuts, legumes, and boron-rich water). Daily dietary intake will be monitored and adjusted to ensure consistent boron exposure.
  Arms: Boron-rich Diet

SUMMARY:
This study investigated the effects of a boron-rich diet compared with a Mediterranean-style diet (Smart Alternative Food Formulation; SAFF) on obesity-related outcomes in adults. Forty obese participants were randomly assigned to receive either a boron-rich diet or the SAFF diet for four weeks. Anthropometric measurements, biochemical parameters, and adipokine levels were evaluated before and after the intervention.

The primary aim was to determine whether dietary boron intake can improve metabolic health, lipid profile, and obesity-related hormonal regulation compared to a widely accepted dietary model. Findings from this trial may contribute to understanding the potential role of boron and diet-microbiota interactions in obesity management and provide evidence for future nutritional strategies.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled clinical trial was conducted to investigate the effects of a boron-rich diet compared to a Mediterranean-style diet (SAFF) on obesity, metabolic parameters, and gut microbiota composition in adults with obesity. The trial was carried out at Dicle University, Diyarbakır, Turkey, over a 4-week intervention period.

A total of 40 obese participants (Body Mass Index [BMI] ≥30 kg/m²), aged 18-65 years, were enrolled following eligibility screening. Inclusion criteria comprised clinically stable individuals without severe systemic disease, no recent antibiotic or probiotic use within the past month, and willingness to comply with dietary instructions. Exclusion criteria included pregnancy or lactation, use of medications affecting weight or metabolism, history of gastrointestinal surgery, or presence of chronic inflammatory diseases.

Participants were randomized into two groups:

Boron-Rich Diet Group (n=20): Participants received a structured diet plan enriched with natural boron sources (such as dried fruits, nuts, legumes, and selected vegetables), formulated to provide a daily boron intake aligned with nutritional safety guidelines.

SAFF (Mediterranean-Style) Diet Group (n=20): Participants followed a diet rich in olive oil, whole grains, legumes, fruits, vegetables, and moderate fish consumption, consistent with Mediterranean dietary principles.

Both groups received equivalent calorie prescriptions tailored to individual energy requirements to promote weight reduction while ensuring comparable macronutrient distribution. Participants received weekly dietary counseling to ensure adherence.

Outcome Measures:

Primary Outcomes: Changes in anthropometric parameters (body weight, BMI, waist circumference) and biochemical markers (lipid profile, fasting glucose, insulin, Homeostatic Model Assessment for Insulin Resistance [HOMA-IR]).

Secondary Outcomes: Serum adipokines (leptin, adiponectin), inflammatory biomarkers, and gut microbiota composition assessed through stool sampling and next-generation sequencing.

Statistical analysis was performed using appropriate parametric or non-parametric tests depending on distribution. Effect sizes and 95% confidence intervals were reported to evaluate the magnitude of differences.

Ethical approval for the study was granted by the Non-Interventional Research Ethics Committee of Firat University (Decision No: 2023/01-19). The trial was conducted in accordance with the principles of the Declaration of Helsinki. Written informed consent was obtained from all participants.

This study contributes novel clinical evidence regarding the potential role of boron-enriched diets as a nutritional intervention for obesity management and provides insights into the diet-microbiota-metabolism relationship.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-65 years
* Body Mass Index (BMI) ≥30 kg/m² (diagnosis of obesity)
* Willingness to participate in the 4-week dietary intervention
* Ability to provide written informed consent

Exclusion Criteria:

* Presence of chronic diseases (e.g., diabetes, cardiovascular disease, renal disease, gastrointestinal disorders)
* Current use of medications or dietary supplements affecting weight, metabolism, or gut microbiota
* Use of probiotics, prebiotics, or commercial weight loss products in the past 3 months
* Pregnancy or lactation
* Known food allergies or intolerances incompatible with the prescribed diets
* Inability to comply with study procedures or dietary intervention

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population is restricted to female participants. Only women who meet the inclusion criteria will be enrolled.
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | Baseline to 4 weeks
  BMI will be calculated as weight (kg) divided by height (m²). Weight will be measured using a calibrated digital scale and height with a stadiometer by trained staff following standardized procedures. The between-group difference in BMI change will be assessed to evaluate the effect of the interventions on obesity outcomes.
Change in Gut Microbiota Diversity | Baseline to 4 weeks
  Stool samples will be collected at baseline and 4 weeks. 16S rRNA gene sequencing will be performed; alpha diversity will be calculated using the Shannon Index. Higher values indicate greater within-sample diversity.

SECONDARY OUTCOMES:
Change in Serum Leptin Level | Baseline to 4 weeks
  Fasting venous blood will be collected in the morning. Serum leptin will be quantified using a validated ELISA kit according to the manufacturer's instructions. Changes will be analyzed within and between diet arms.
Change in Low-Density Lipoprotein Cholesterol | Baseline to 4 weeks
  Fasting lipid profile will be measured using an automated analyzer in the central laboratory. LDL-C will be calculated directly or via the Friedewald equation when applicable. The outcome represents the change in LDL-C from baseline to end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Feray Çağıran Yılmaz, Associate Professor, Principal, Principal Investigator — Dicle Üniversitesi
Locations (1):
- Feray Çağıran Yılmaz, Diyarbakır, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No